CLINICAL TRIAL: NCT03073044
Title: Italian Validation of the Belastungfragebogen Parkinson Kurzversion (BELA-P-K): a Disease-specific Questionnaire for Evaluation of the Subjective Perception of Quality of Life.
Brief Title: Translation and Validation of BELA-p-K for QoL Evaluation in PD Patients
Status: Completed | Type: Observational
Sponsor: Ospedale Generale Di Zona Moriggia-Pelascini (Other)
Responsible Party: Principal Investigator, Ilaria Zivi, Dipartimento di riabilitazione malattia di Parkinson, Disturbi del movimento e Cerebrolesioni Acquisite, Ospedale Generale Di Zona Moriggia-Pelascini
Other Study IDs: Bela-p-K
Record Dates: First submitted 2017-02-22; First posted 2017-03-08 (Actual); Last update posted 2017-03-08 (Actual); Status verified 2017-03

CONDITIONS: Parkinson Disease
Keywords: Quality of life; psychosocial and psychological problems
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: BELASTUNGSFRAGEBOGEN PARKINSON KURZVERSION (BELA-P-K) — we proposed the translation and validation of Bela-p-K, a questionnaire that evaluates the Quality of Life in parkinsonian patients.
  we applied the method of translation and back-translation at dutch version of questionnaire. after, we evaluated 103 PD patients with Bela-p-K and PDQ39.
  The internal consistency of questionnaire was analyzed calculating alpha-Chronbach. We also evaluated the construct validity correlating Bela-p-K and PDQ39

SUMMARY:
The BELA-P-k was translated from Dutch into Italian. Subsequently 102 patients with PD filled out the questionnaire

DETAILED DESCRIPTION:
In order to provide an appropriate endpoint for the assessment of the effectiveness of rehabilitation treatments on QoL of PD patients, in this study we translated and then validated the Belastungsfragebogen Parkinson kurzversion (BELA-P-k). This tool allows evaluating separately two crucial aspects: i) the loss of personal autonomy in activities of daily life and ii) the psychological and psychosocial impact of the disease.

The BELA-P-k was translated from Dutch into Italian. Subsequently 102 patients with PD filled out the questionnaire. PD patients were also evaluated by using the Parkinson Disease Questionnaire -39 (PDQ39), the Unified Parkinson's Disease Rating Scale (UPDRS), the Mini Mental State Examination (MMSE) and the Frontal Assessment Battery (FAB) The internal consistency of the questionnaire was assessed by means of Cronbach's alpha coefficient.

The discriminant validity was assessed by testing for differences between mean values for patients grouped according to Hoehn and Yahr stages. This analysis was carried out by a one-way analysis of variance.

Finally, the construct validity was determined by assessing the relationship (Spearman rank correlation coefficient) between Bela-P-k and the PDQ39

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's Disease

Exclusion Criteria:

* any focal brain lesion detected in brain imaging studies (CT or MRI) performed in the previous twelve months;
* other chronic diseases with a known impact in QoL.
* MMSE < 24

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with idiopathic Parkinson Disease
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Bela-p-K | 15 minuts
  questionnaire for QoL evaluation

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spliethoff-Kamminga NG, Zwinderman AH, Springer MP, Roos RA. Psychosocial problems in Parkinson's disease: evaluation of a disease-specific questionnaire. Mov Disord. 2003 May;18(5):503-9. doi: 10.1002/mds.10388. PMID 12722163
- [Background] Ringendahl H, Werheid K, Leplow B, Ellgring H, Annecke R, Emmans D. [Recommendations for standarsized psychological diagnosis in Parkinson patients]. Nervenarzt. 2000 Dec;71(12):946-54. doi: 10.1007/s001150050691. German. PMID 11139990
- [Derived] Ortelli P, Maestri R, Zarucchi M, Cian V, Urso E, Giacomello F, Ferrazzoli D, Frazzitta G. Italian validation of the Belastungsfragebogen Parkinson kurzversion (BELA-P-k): a disease-specific questionnaire for evaluation of the subjective perception of quality of life in parkinson's disease. J Clin Mov Disord. 2017 Jul 25;4:12. doi: 10.1186/s40734-017-0059-x. eCollection 2017. PMID 28770096